CLINICAL TRIAL: NCT01657357
Title: Routine Follow up After THA in PAO Patient
Brief Title: Routine Follow up After Total Hip Arthroplasty Prior Periacetabular Osteotomy
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: THA after PAO
Record Dates: First submitted 2012-03-13; First posted 2012-08-06 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Hip Dysplasia; Osteotomy of Pelvis; Total Hip Arthroplasty
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PAO, osteoarhritis, THA
  Interventions: Other: Routine followup

INTERVENTIONS:
Other: Routine followup — questionnaires

SUMMARY:
Follow up study of patients, who despite periacetabular osteotomy, need a total hip arthroplasty, to see outcome.

ELIGIBILITY:
Inclusion Criteria:

* PAO and THA

Exclusion Criteria:

* time since THA less than 4 yrs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, who despite a joint preserving procedure(periacetabular osteotomy PAO) ended up with a total hip arthroplasty (THA).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Does previous PAO compromise the function of a secondary THA | Up to 10 years after THA surgery
  To describe the radiographic status (ex. cup positioning, calcifications, signs of loosing etc) of the THA, the physical function of the THA ( Harris Hip Score), and pt reported outcome measurements (SF36 and WOMAC).

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Prof. D.Msc, Study Chair — Orthopedic Research Unit, Aarhus University Hospital; Charlotte Hartig-Andreasen, MD, Principal Investigator — Orthopedic Research Unit, Aarhus University Hospital
Locations (1):
- Orthopaedic department, Aarhus Universityhospital, Aarhus, Aarhus, Denmark